CLINICAL TRIAL: NCT01071018
Title: A Phase I Study of MK2206 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of MK2206 in Locally Advanced or Metastatic Solid Tumors (2206-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2206-007; 2010_509
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Solid Tumors
Keywords: locally advanced or metastatic solid tumors
MeSH Terms: interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- QOD Schedule (Experimental): QOD Schedule, MK2206 every other day
  Interventions: Drug: MK2206 every other day
- QW Schedule (Experimental): QW Schedule, MK2206 once weekly
  Interventions: Drug: MK2206 once weekly

INTERVENTIONS:
Drug: MK2206 every other day — Dose escalation study: MK2206 will be administered as an oral formulation in rising dose levels of 45 mg and 60 mg, once daily every other day in repeating 4 week cycles.
  Other Names: MK2206
  Arms: QOD Schedule
Drug: MK2206 once weekly — Dose escalation study: MK2206 will be administered as an oral formulation in rising dose levels of 135 mg and 200 mg, once weekly in repeating 4 week cycles.
  Other Names: MK2206
  Arms: QW Schedule

SUMMARY:
This study is designed to evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics and anti-tumor activity of MK2206 when administered with Every Other Day (QOD) and Once Weekly (QW) dosing schedules.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have confirmed locally advanced or metastatic solid tumors that have failed to respond to standard therapy, have gotten worse or have come back after existing therapy
* Has adequate organ function
* Is ECOG Performance Scale 0-1
* Has a negative urine pregnancy test if patient is female
* Is able to swallow capsules and has no surgical or bodily condition that will prevent the patient from swallowing and absorbing oral medications on an ongoing basis

Exclusion Criteria:

* Patient has had chemotherapy, radiotherapy, biological therapy or surgery within 4 weeks of starting the study and has not recovered from adverse events caused by the treatment
* Is currently participating or has participated in a study with an investigational compound or device within 28 days
* Has a primary central nervous system tumor
* Has a history or current evidence of heart disease, slow heart rate or untreated high blood pressure
* Is a known diabetic who is taking insulin or oral antidiabetic therapy
* Is pregnant or breastfeeding or planning to become pregnant during the study
* Is positive HIV antibody, HBs antigen or HCV antibody

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Characterize safety and tolerability of MK2206 by monitoring incidence of protocol-defined dose limiting toxicities (DLTs) | Day 1 - Day 28 (Cycle 1)

SECONDARY OUTCOMES:
Assess pharmacokinetic (PK) profile of MK2206 by determining parameters: AUC, Cmax, and Tmax | Day 1 - Day 28 (Cycle 1)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Doi T, Tamura K, Tanabe Y, Yonemori K, Yoshino T, Fuse N, Kodaira M, Bando H, Noguchi K, Shimamoto T, Ohtsu A. Phase 1 pharmacokinetic study of the oral pan-AKT inhibitor MK-2206 in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2015 Aug;76(2):409-16. doi: 10.1007/s00280-015-2810-z. Epub 2015 Jun 24. PMID 26104654